CLINICAL TRIAL: NCT02531646
Title: Clinical Evaluation of CARESTREAM Dual Energy and Digital Tomosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 9J8068
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2015-08

CONDITIONS: Solitary Pulmonary Nodules
Keywords: pulmonary nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Predicate & Invest. DE - Human Subjects (Experimental): Radiation -Thirty to forty (30-40) patients will receive a DR standard of care chest exam using the DRX Plus detector and a DE exam. Each DE patient exam includes high energy and low energy image exposures using the investigational device. These images are used by the DE console software to generate additional DE images (e.g. bone and soft tissue).
  Interventions: Radiation: Radiation
- Predicate & Invest. DT - Human Subjects (Experimental): Radiation - Fifteen to twenty (15-20) patients will receive a DR standard of care chest exam using the DRX Plus detector, and a DT exam. Each DT patient exam includes a scout image (chest PA) and a DT scan using the investigational DT SW. The DT scan is used by the DT console software to generate tomographic images.
  Interventions: Radiation: Radiation
- Predicate & Invest. DT - Phantom Images (Experimental): Radiation - Eleven (11) phantoms of various anatomy will be imaged with linear tomography (LT) as predicate and DT for investigational.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation - Each human subject will receive one standard of care x-ray and one Duel Energy exposure or one standard of care x-ray and one Digital Tomosynthesis exposure. Phantoms were imaged using linear tomography and digital tomography.

SUMMARY:
The purpose of this study is to evaluate the imaging performance of Dual Energy and Digital Tomosynthesis (DE-DT) application against the commercially available predicate devices.

DETAILED DESCRIPTION:
The acquisition system will consist of using site equipment including the CARESTREAM DRX-Evolution x-ray system, and the predicate CARESTREAM DRX Plus detector and the investigational DE-DT application.

DE Study Design Thirty to forty (30-40) patients will receive a DR standard of care chest exam using the DRX Plus detector and a DE exam. Each DE patient exam includes high energy and low energy image exposures using the investigational device. These images are used by the DE console software to generate additional DE images (e.g. bone and soft tissue).

DT Study Design Fifteen to twenty (15-20) patients will receive a DR standard of care chest exam using the DRX Plus detector, and a DT exam. Each DT patient exam includes a scout image (chest PA) and a DT scan using the investigational DT SW. The DT scan is used by the DT console software to generate tomographic images.

11 phantoms of various anatomy will be imaged with linear tomography (LT) as predicate and DT for investigational.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years and older. Subject has provided informed consent. Study participant is scheduled to have a chest CT exam. Study participant is able to stand and be still during the exams.

Exclusion Criteria:

Human subject specific:

Not able or willing to provide Informed Consent, or consent is withdrawn. Study participant is a female of child bearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, MD, Principal Investigator — Toronto General Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Predicate & Invest. DE - Human Subjects: Radiation -Thirty to forty (30-40) patients will receive a DR standard of care chest exam using the DRX Plus detector and a DE exam. Each DE patient exam includes high energy and low energy image exposures using the investigational device. These images are used by the DE console software to generate additional DE images (e.g. bone and soft tissue).
  Radiation: Radiation - Each human subject will receive one standard of care x-ray and one Duel Energy exposure or one standard of care x-ray and one Digital Tomosynthesis exposure.
- Predicate & Invest. DT - Human Subjects: Radiation - Fifteen to twenty (15-20) patients will receive a DR standard of care chest exam using the DRX Plus detector, and a DT exam. Each DT patient exam includes a scout image (chest PA) and a DT scan using the investigational DT SW. The DT scan is used by the DT console software to generate tomographic images.
  Radiation: Radiation - Each human subject will receive one standard of care x-ray and one Duel Energy exposure or one standard of care x-ray and one Digital Tomosynthesis exposure.
- Predicate & Invest. DT - Phantom Images: Radiation - Eleven (11) phantoms of various anatomy will be imaged with linear tomography (LT) as predicate and DT for investigational.
  Radiation: Radiation - Each human subject will receive one standard of care x-ray and one Duel Energy exposure or one standard of care x-ray and one Digital Tomosynthesis exposure.
Period: Overall Study
Arm/Group | Predicate & Invest. DE - Human Subjects | Predicate & Invest. DT - Human Subjects | Predicate & Invest. DT - Phantom Images
Started | 37 | 18 | 11
Completed | 32 | 17 | 11
Not Completed | 5 | 1 | 0
Not completed — equip. image processing issue | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 37 live human DE cases, 18 live human DT cases, 11 phantom images.
Groups:
- Total: Total of all reporting groups
Arm/Group | Predicate & Invest. DE - Human Subjects | Predicate & Invest. DT - Human Subjects | Predicate & Invest. DT - Phantom Images | Total
Number analyzed (Participants) | 37 | 18 | 11 | 66
Age, Customized [Number; unit: years]
  > 18 years | 37 | 18 | 11 | 66
Sex/Gender, Customized [Number; unit: participants]
  unknown | 37 | 18 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DE Predicate PA Chest
Description: 1-1.9-Non-diagnostic Unacceptable for diagnostic purposes. Little or no clinically usable diagnostic information (e.g., gross underexposure, system failure or extensive motion artifact). Almost all such imaging should be repeated. 2-2.9-Limited Acceptable, with some technical defect (motion artifact, body habitus/poor x-ray penetration, or patient positioning may limit visualization of some body-regions but still adequate for diagnostic purposes). Not as much diagnostic information as is typical for an examination of this type, but likely sufficient. 3-3.9-Diagnostic Image quality that would be expected routinely when imaging cooperative patients. 4-Exemplary Good, most adequate for diagnostic purposes. Image quality that can serve as an example that should be emulated.
Time Frame: 3 months
Population: 224 image ratings from 7 radiologist readers (32 images rated x 7 readers) for Predicate & Invest. DE - Human Subjects arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DE - Human Subjects
Number analyzed (Participants) | 32
Number analyzed (images) | 224
units on a scale | 3.4540 (0.0183)

2. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DE Investigational Composite
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DE - Human Subjects
Number analyzed (Participants) | 32
Number analyzed (images) | 224
units on a scale | 3.3214 (0.0242)
Statistical Analysis 1: Comparison: Predicate & Invest. DE - Human Subjects; Test type: Non-Inferiority or Equivalence — Equivalence interval (-0.25, 0.25); p = 0.000, Equivalence test — Level of significance (alpha) = 0.05 All p-values were calculated (and verified) by our statistician.They were rounded to fit four digits

3. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DE Investigational High Energy
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DE - Human Subjects
Number analyzed (Participants) | 32
Number analyzed (images) | 224
units on a scale | 3.2911 (0.0178)
Statistical Analysis 1: Comparison: Predicate & Invest. DE - Human Subjects; Test type: Non-Inferiority or Equivalence — Equivalence interval (-0.25, 0.25); p = 0.000, Equivalence test — [p-value comment as in outcome 2, analysis 1]

4. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DE Investigational Low Energy
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DE - Human Subjects
Number analyzed (Participants) | 32
Number analyzed (images) | 224
units on a scale | 3.5504 (0.0163)
Statistical Analysis 1: Comparison: Predicate & Invest. DE - Human Subjects; Test type: Superiority or Other; p = 0.000, t-test, 1 sided — [p-value comment as in outcome 2, analysis 1]

5. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DT Reference 1- PA Chest
Description: as for outcome 1
Time Frame: 3 months
Population: 119 image ratings from 7 radiologist readers (17 images rated x 7 readers) for Predicate & Invest. DT Reference 1 - PA Chest arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DT - Human Subjects
Number analyzed (Participants) | 17
Number analyzed (images) | 119
units on a scale | 3.4832 (0.0228)
Statistical Analysis 1: Comparison: Predicate & Invest. DT - Human Subjects; Test type: Superiority or Other; p = 0.000, t-test, 1 sided — Level of significance (alpha) = 0.05 All p-values were calculated (and verified) by our statistician. They were rounded to fit four digits

6. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DT Reference 2 - PA and LAT Chest
Description: as for outcome 1
Time Frame: 3 months
Population: 119 image ratings from 7 radiologist readers (17 images rated x 7 readers) for Predicate & Invest. DT Reference 2 - PA and LAT Chest arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DT - Human Subjects
Number analyzed (Participants) | 17
Number analyzed (images) | 119
units on a scale | 3.5546 (0.0190)
Statistical Analysis 1: Comparison: Predicate & Invest. DT - Human Subjects; Test type: Superiority or Other; p = 0.007, t-test, 1 sided — [p-value comment as in outcome 5, analysis 1]

7. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DT Investigational - Scout & DT Volume
Description: as for outcome 1
Time Frame: 3 month
Population: 119 image ratings from 7 radiologist readers (17 images rated x 7 readers) for DT Investigational - Scout & DT Volume.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DT - Human Subjects
Number analyzed (Participants) | 17
Number analyzed (images) | 119
units on a scale | 3.6277 (0.0230)

8. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - LT Predicate Phantom Images
Description: as for outcome 1
Time Frame: 3 months
Population: 77 phantom image ratings from 7 radiologist readers (11 images rated x 7 readers) for Predicate & Invest. DT - Phantom Images arm above.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DT - Phantom Images
Number analyzed (Participants) | 11
Number analyzed (images) | 77
units on a scale | 3.3494 (0.0433)
Statistical Analysis 1: Comparison: Predicate & Invest. DT - Phantom Images; Test type: Superiority or Other; p = 0.000, t-test, 1 sided — [p-value comment as in outcome 5, analysis 1]

9. Primary Outcome: Radlex Scale for Diagnostic Quality Ratings - DT Investigational Phantom Images
Description: as for outcome 1
Time Frame: 3 months
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: images
Arm/Group | Predicate & Invest. DT - Phantom Images
Number analyzed (Participants) | 11
Number analyzed (images) | 77
units on a scale | 3.7156 (0.0268)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Predicate & Invest. DE - Human Subjects | Predicate & Invest. DT - Human Subjects | Predicate & Invest. DT - Phantom Images
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/32 | 0/17 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No